CLINICAL TRIAL: NCT03755817
Title: Immediate Efficacy Assessment of SCENAR's Session on a Common Spinal Pain Syndrome
Brief Title: Efficacy Assessment of SCENAR Device on Common Spinal Pain Syndrome
Acronym: SCENAR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017015F
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pain Syndrome
Keywords: Spinal pain
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scenar application (Experimental): Application of SCENAR device on
  Interventions: Device: SCENAR application
- Scenar application with the device off (Placebo Comparator): Application of SCENAR device off
  Interventions: Device: SCENAR application with the device off

INTERVENTIONS:
Device: SCENAR application — Active SCENAR application on the painful area
  Arms: Scenar application
Device: SCENAR application with the device off — Placebo SCENAR application on the painful area
  Arms: Scenar application with the device off

SUMMARY:
Randomized, singled blinded, controlled trial of the efficacy of a SCENAR session in patients with vertebral pain. SCENAR is an electrotherapy device.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 and under 80 years of age
* Suffering of common spinal pain: cervical pain including cervico-brachial neuralgia, lumbar pain including lumbo-radiculalgia
* Having attended a "pain consultation" or referred to a pain consultant during hospitalization
* Having signed the consent form
* Can be contacted directly by phone if patient is not hospitalized
* Be affiliated to a national insurance scheme or benefiting from such a program

Non-inclusion Criteria:

* Pregnant or breast-feeding women
* Patients with a pacemaker
* Patients whose skin condition makes the use of SCENAR impossible (wounds, recent scars, skin infections)
* Patient whose spinal pain is known to be related to inflammatory pathology (spondylarthropathy, rheumatoid arthritis, chondrocalcinosis), trauma (fractures and dislocations), tumor (metastases, myeloma localization), spondylodiscitis infectious, neurological (intrarachidian tumor or posterior fossa) or radiculalgia with deficient signs
* Patients who have already had a SCENAR session
* Patients who have already participated in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Efficacy on resting pain at the end of SCENAR application: NRS | 30 minutes
  Self-assessment of pain using the pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain")

SECONDARY OUTCOMES:
Efficacy on pain at mobilization the end of SCENAR application: NRS | 30 minutes
  Self-assessment of pain intensity using the pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain")
Efficacy on anxiety the end of SCENAR application: NRS | 30 minutes
  Self-assessment of anxiety using the pain numeric rating scale (NRS), on which patients rate their current anxiety from 0 ("no anxiety") to 10 ("worst possible anxiety")
Efficacy on the sensation of spinal blockage at the end of SCENAR application: NRS | 30 minutes
  Self-assessment of the sensation of spinal blockage using the numeric rating scale (NRS), on which patients rate their current blockage from 0 ("complete blockage") to 10 ("perfect mobility")
Efficacy on resting pain on the following day: NRS | 1 day
  Self-assessment of pain using the pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain")
Efficacy on pain at mobilization on the following day: NRS | 1 day
  Self-assessment of pain using the pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain")
Efficacy on the sensation of spinal blockage on the following day: NRS | 1 day
  Self-assessment of the sensation of spinal blockage using the numeric rating scale (NRS), on which patients rate their current anxiety from 0 ("complete blockage") to 10 ("perfect mobility")
Efficacy on anxiety on the following day: NRS | 1 day
  Self-assessment of anxiety using the numeric rating scale (NRS), on which patients rate their current anxiety from 0 ("no anxiety") to 10 ("worst possible anxiety")
Collection of possible side effects | 1 day
  Open question

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD PhD, Study Director — Hopital Foch
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No